CLINICAL TRIAL: NCT03179579
Title: A Phase III Study of Hyperthermic Intraperitoneal Chemotherapy (HIPEC) Combined With Systemic Chemotherapy And Cytoreductive Surgery (CRS) in the Treatment of Peritoneal Carcinomatosis From Gastric Cancer
Brief Title: Efficacy of HIPEC Combined With Systemic Chemotherapy and CRS on Peritoneal Metastases From Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shu-Zhong Cui (Other)
Collaborators: Tianjin Medical University Cancer Institute and Hospital (Other); Chinese PLA General Hospital (Other); Harbin Medical University (Other); Southern Medical University, China (Other); Guangdong Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Shu-Zhong Cui, President of Affiliated Tumor Hospital of Guangzhou Medical, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Organization: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIPEC-02
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Gastric Cancer; Peritoneal Carcinomatosis
Keywords: Gastric Cancer; Peritoneal Carcinomatosis; Hyperthermic Intraperitoneal Chemotherapy; Systemic Chemotherapy; Cytoreductive Surgery
MeSH Terms: conditions — Stomach Neoplasms; Peritoneal Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 1. HIPEC with paclitaxel 135 mg/m^2+HIPEC with cisplatin 75 mg/m^2±HIPEC with Raltitrexed 3 mg/m^2 intraperitoneally in succession
  2. 2 cycles of neoadjuvant chemotherapy: S-1 40-60 mg/m^2, d1-d14, Bid p.o.+ oxaliplatin 130 mg/m^2, d1, IV, every 3 weeks
  3. Cytoreductive surgery
  4. HIPEC with paclitaxel 135 mg/m^2+HIPEC with cisplatin 75 mg/m^2±HIPEC with Raltitrexed 3 mg/m^2 intraperitoneally in succession
  5. 4-6 cycles of adjuvant chemotherapy: S-1 40-60 mg/m^2, d1-d14, Bid p.o.+ oxaliplatin 130 mg/m^2, d1, IV, every 3 weeks
  Interventions: Procedure: HIPEC with neoadjuvant chemotherapy
- Control group (Active Comparator): 1. 3 cycles of neoadjuvant chemotherapy: S-1 40-60 mg/m^2, d1-d14, Bid p.o.+ oxaliplatin 130 mg/m^2, d1, IV, every 3 weeks
  2. Cytoreductive surgery
  3. 4-6 cycles of adjuvant chemotherapy: S-1 40-60 mg/m^2, d1-d14, Bid p.o.+ oxaliplatin 130 mg/m^2, d1, IV, every 3 weeks
  Interventions: Procedure: Systemic chemotherapy

INTERVENTIONS:
Procedure: HIPEC with neoadjuvant chemotherapy — HIPEC 3 times +NACT 2 cycles +CRS +HIPEC 3 times+ ACT 4-6 cycles
  Other Names: CRS with HIPEC and adjuvant cheomtherapy
  Arms: Experimental group
Procedure: Systemic chemotherapy — NACT 3 cycles +CRS +ACT 4-6 cycles
  Other Names: CRS with systemic chemotherpay
  Arms: Control group

SUMMARY:
This project is a multi-center, prospective, randomized controlled clinical observation the safety and efficacy that stage IV limited peritoneal metastasis of gastric cancer patients accept hyperthermic intraperitoneal chemotherapy plus neoadjuvant chemotherapy with CRS and systemic chemotherapy. With advanced-stage gastric patients of confined to the peritoneal as the research object, with median progression-free survival and overall survival, adverse events as the end points.

DETAILED DESCRIPTION:
Peritoneal metastases in gastric cancer are considered as terminal disease with poor prognosis, the median survival time of this kind of patients is less than 1 year and even worse in China. Recently, cytoreductive surgery (CRS) combined with hyperthermic intraperitoneal chemotherapy (HIPEC) has been suggested to improve survival in patients with peritoneal metastases from gastric cancer. Even though the REGATTA trial demonstrated that the removal of the primary tumor is not necessarily beneficial, the role of operation aiming at R0 resection combined with new regimens like HIPEC and new chemotherapeutic agents is still confusing. Neoadjuvant chemotherapy prolonged OS of patients received macroscopically radical (CC0) surgery. Compared to systemic chemotherapy, HIPEC promotes chemotherapy to penetrate deeper into the cancer tissue, which needed multicenter randomized clinical trials (RCTs) to comfirm. Therefore, we has conducting prospective phase III trial of HIPEC combined with systemic chemotherapy and CRS for gastric cancer with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Gastic adenocarcinoma is diagnosed by histological and cytological examination.
2. Peritoneal carcinomastosis of gastric cancer is diagnosed by laparotomy or laparoscopic exploration.
3. According to Sugarbaker's peritoneal cancer index (PCI), PCI score of participant is no more than 20.
4. 18 < Age < 70 year old
5. Expected survival > 3 months
6. Performance status: ECOG 0-1
7. Adequate bone marrow function Hb ≥9 g/dl (After correction in case of iron deficient anemia) WBC ≥ 3,500/mm3, Platelet ≥ 100,000/mm3
8. Adequate renal function Creatinine ≤ 1.5 mg/dl, and adequate hepatic function Bilirubin ≤ 1.5 mg/dl and AST and ALT ≤ 2.5×ULN

10. Voluntary participation after getting written informed consent.

Exclusion Criteria:

1. Except for peritoneal carcinomatosis, gastric cancer concurrently metastasized to liver, lung, para-aortic lymph node and other distant organs.
2. Extensive adhesion in peritoneal cavity
3. Previous History of other malignancies
4. Poorly controlled disease e.g. atrial fibrillation, stenocardia, cardiac insufficiency, persistent hypertension despite medicinal treatment, ejection fraction<50%
5. Receiving other chemotherapy, radiotherapy or immunotherapy
6. Patients who are unsuitable candidates by doctor's decision
7. Without given written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Median overall survival | 3 years
  assess median overall survival rate during 3 years in both study arms

SECONDARY OUTCOMES:
Risk factors for morbidity and mortality | Through study completion, an average of 1 year.
  determine percent of patients wtih Grade I-IV adverse events according to NCI criteria, Common Terminology Criteria for AE (CTCAE 4.0).

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Zhong Cui, M.D, Study Chair — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Department of Abdominal Surgery (Section 2), Affiliated Tumor Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No